CLINICAL TRIAL: NCT01928953
Title: Longitudinal Study of Patients With Opioid-Induced Constipation
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: 12AST11894/A-12292
Record Dates: First submitted 2013-08-22; First posted 2013-08-27 (Estimated); Last update posted 2015-07-08 (Estimated); Status verified 2015-07

CONDITIONS: Patients With Opioid Induced Constipation
Keywords: opioid induced constipation in patients without cancer and with cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This prospective hybrid longitudinal study was conducted in the United States (US), Canada, the United Kingdom (UK), and Germany. To obtain the most complete and comprehensive understanding of the burden of opioid-induced constipation (OIC) in these countries, this study used a combination of web-based, longitudinal patient survey, retrospective data abstraction from medical records, and a prospective physician survey.

The primary objective of this study was to estimate the rate of inadequate response to laxatives (LIR), which was defined as having sufficient laxative use (at least one laxative use ≥ four times per reference period), and inadequate response (defined as fewer than three bowel movements (BMs) OR at least one of the following symptoms on the Patient Assessment of Constipation Symptoms (PAC-SYM) measure scored as moderate, severe or very severe: BMs too hard, straining to have a BM, feeling like you didn't "finish" a BM, and feeling like you had to pass a BM but could not), in a cohort of non-cancer pain and cancer pain (separately) participants with OIC, by country and overall.

The secondary study objectives are as follows:

1. To estimate the rate of LIR for two subgroups: 1xLIR and 2xLIR. 1xLIR was defined as use of at least one laxative agent ≥ 4 times in the reference period while 2xLIR was defined as the use of at least two laxative agents, each used ≥ 4 times in the reference period;
2. To describe the baseline demographic and clinical characteristics, including prior health status, comorbidities, constipation-related GI symptoms, and concomitant medications of patients with OIC;
3. To describe drug utilization and self-management of OIC;
4. To describe the pre-index and post-index healthcare resource utilization and estimate costs associated with the diagnosis, treatment, and general management of OIC (including laxative use) and events attributed to OIC, including both direct and indirect costs;
5. To describe patient-reported impact of OIC on health-related quality of life, productivity, and pain management;
6. To describe patient-reported treatment satisfaction with laxative use; and
7. To describe physician-reported awareness of OIC and symptoms and understanding of patient-reported impact of OIC.

ELIGIBILITY:
Inclusion Criteria:

* Patient is receiving a minimum total daily dose of 30 mg of oral morphine, or equianalgesic amount[s] of 1 or more other opioid therapies, for a minimum of 4 weeks for chronic pain or cancer relate pain Presence of OIC in the past 2 weeks

  * (for cancer patients only) Patient has a current diagnosis of cancer that is not currently in remission and has cancer-related pain Internet access and is able and willing to complete a longitudinal web-based survey
  * Patient is able to understand and comply with the requirements of the study, as judged by the investigator (includes ability to read and write and to use

Exclusion Criteria:

* Patient is unable or refuses to provide informed consent;

  * Patient does not have access to a computer with internet connectivity, or is unable to use a computer to complete the web-based survey; Based on clinical judgment, patient has a history of chronic constipation (i.e. clinical diagnosis, note in the medical record, or patient history);
  * Patient has a history of (or current) colon cancer (primary or metastatic) (i.e., clinical diagnosis Patient has received an investigational medication to treat constipation or participated in any study involving investigational compound naloxegol within ≤90 days prior to the baseline visit

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population consists of patients who have been on daily opioid therapy for ≥ 4 weeks for the treatment of chronic non-cancer or cancer pain and who have opioid-induced constipation, as per patient history.
Sampling Method: Probability Sample
Enrollment: 520 (Actual)
Dates: Start 2012-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Rate of LIR among the OIC population | 6 months

SECONDARY OUTCOMES:
Rate of inadequate response to first and second-line laxative treatment for OIC (1x LIR and 2x LIR). | 6 months
Baseline demographic and clinical characteristics of patients with OIC (prior health status, comorbidities, GI symptoms, and concomitant medications). | 12months retrospectively
Drug utilization and self-management of OIC at baseline and changes from baseline over the 24-week follow-up period. | 6 months
Healthcare resource utilization profiles pre- and post-baseline | 6 months
Cost of illness related to the diagnosis, treatment, and general management of OIC (including laxative use) and events attributed to OIC, including both direct and indirect costs. | 6 months
Baseline constipation-associated GI symptoms and changes from baseline over the 24-week follow-up period (PAC-SYM and additional symptom questions). | 6 months
Baseline health-related quality of life (PAC-QOL and EQ-5D) and changes from baseline over the 24-week follow-up period (PAC-QOL). | 6 months
Loss of productivity (WPAI-SHP score) at baseline and changes from baseline over the 24-week follow-up period. | 6 months
Persistence on opioid therapy at baseline and changes from baseline over the 24-week follow-up period | 6 months
Treatment satisfaction with laxative use at baseline and changes from baseline over the 24-week follow-up period, for all patients taking laxatives. | 6 months
Physician-reported awareness of OIC and symptoms, and understanding of patient reported impact of OIC at baseline. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Mark Sostek, M.D., Study Director — AstraZeneca; Cathy Datto, M.D., M.S., Study Director — AstraZeneca; Robert J LoCasale, Phd, MS, Principal Investigator — AstraZeneca
Locations (30):
- United States (24):
  - Alliance Clinical Research, Birmingham, Alabama
  - Horizon Research Group, Inc, Mobile, Alabama
  - HOPE Research Institute, Phoenix, Arizona
  - Advanced Rx Clinical Research, Artelia, California
  - TriWest Research Associates, LLC, El Cajon, California
  - Akkiance Research Centers, Laguna Hills, California
  - Primecare Clinical Research, Lajuna Hills, California
  - Samaritan Center for Medical Research, Los Gatos, California
  - Precision Research Institute, LLC, San Diego, California
  - Southeast Clinical Research, LLC, Jacksonville, Florida
  - Physician Care Clinical Research, LLC, Sarasota, Florida
  - Soth Miami Clinical Research, South Miami, Florida
  - Chicago Anesthesia Pain Specialists, Chicago, Illinois
  - ActivMed Practices & Research, Newington, New Hampshire
  - Atco Medical Associates, P.C., Atco, New Jersey
  - DiGiovanna Institute for medical Education and Research, North Massapequa, New York
  - Gaffnew Health Services, Charlotte, North Carolina
  - Clinical Inquest Center LTD, Beavercreek, Ohio
  - Ohio Clinical Research Partners, LLC, Canton, Ohio
  - Clinical Inquest Center, Ltd., Dayton, Ohio
  - NPC Research, Oklahoma City, Oklahoma
  - Pain Research of Charleston, Charleston, South Carolina
  - Family Medicine of SayeBrook, Myrtle Beach, South Carolina
  - Highland Clinical Research, Salt Lake City, Utah
- Canada (6):
  - University of Calgary, Calgary, Alberta
  - Paradise Medical Clinic, Paradise, Newfoundland and Labrador
  - Aviva Clinical Trial Group Inc., Burlington, Ontario
  - SKDS Research Inc., Newmarket, Ontario
  - Taunton Health Centre, Oshawa, Ontario
  - Pro-Recherche, Saint Romuald, Quebec

REFERENCES:
- [Derived] Gupta A, Coyne KS, Datto C, Venuti C. The Burden of Opioid-Induced Constipation in Younger Patients with Chronic Noncancer Pain. Pain Med. 2018 Dec 1;19(12):2459-2468. doi: 10.1093/pm/pny002. PMID 29420795
- [Derived] LoCasale RJ, Datto C, Wilson H, Yeomans K, Coyne KS. The Burden of Opioid-Induced Constipation: Discordance Between Patient and Health Care Provider Reports. J Manag Care Spec Pharm. 2016 Mar;22(3):236-45. doi: 10.18553/jmcp.2016.22.3.236. PMID 27003553